CLINICAL TRIAL: NCT01614457
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Ivacaftor in Subjects With Cystic Fibrosis Who Have the R117H-CFTR Mutation
Brief Title: Study of Ivacaftor in Subjects With Cystic Fibrosis (CF) Who Have the R117H-CF Transmembrane Conductance Regulator (CFTR) Mutation (KONDUCT)
Acronym: KONDUCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX11-770-110
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivacaftor (Experimental): Ivacaftor 150 milligram (mg) tablet orally twice daily for 24 weeks.
  Interventions: Drug: Ivacaftor
- Placebo (Placebo Comparator): Placebo matched to Ivacaftor tablet orally twice daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivacaftor — Ivacaftor 150 milligram (mg) tablet orally twice daily for 24 weeks.
  Other Names: Kalydeco; VX-770
  Arms: Ivacaftor
Drug: Placebo — Placebo matched to Ivacaftor tablet orally twice daily for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ivacaftor in subjects with cystic fibrosis (CF) who have the R117H-CFTR mutation.

DETAILED DESCRIPTION:
Ivacaftor is the first CFTR modulator to show an improvement in CFTR function and clinical benefit in subjects with CF. Results from Phase 3 studies (VX08-770-102 [Study 102] [NCT00909532] and VX08-770-103 [Study 103] [NCT00909727]) showed that ivacaftor is effective in the treatment of subjects with CF who have the G551D-CFTR mutation, as evidenced by sustained improvements in CFTR channel function (measured by reduction in sweat chloride concentration) and corresponding substantial, durable improvements in lung function, pulmonary exacerbations, respiratory symptoms, and weight gain. Ivacaftor was also well tolerated, as evidenced by the rates and reasons for premature discontinuation and results of safety assessments.

Ivacaftor (Trade Name Kalydeco; 150 mg tablets) was initially approved in the United States for the treatment of CF in subjects 6 years of age and older who have a G551D mutation in the CFTR gene.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF
* Must have at least 1 allele of the R117H CFTR mutation
* Percent predicted forced expiratory volume in 1 second (FEV1) 40 percent (%) to 90% (for subjects aged 12 years or older) or 40% to 105% (for subjects aged 6 to 11 years) predicted normal for age, sex, and height
* 6 years of age or older
* Minimum weight of 15 kilogram (kg) at screening
* Females of childbearing potential must not be pregnant
* Willing to comply with contraception requirements

Exclusion Criteria:

* CFTR gene mutation leading to CFTR channel with gating defect (that is, any 1 of the following mutations: G551D, G178R, G551S, S549N, S549R, G970R, G1244E, S1251N, S1255P, or G1349D)
* History of any illness or condition that might confound the results of the study or pose an additional risk in administering ivacaftor to the subject
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before the first dose of study drug
* Abnormal liver function, at screening, defined as greater than or equal to (>=) 3 time upper limit of normal (ULN), of any 3 or more of the following: serum aspartate transaminase (AST), serum alanine transaminase (ALT), gamma-glutamyl transpeptidase (GGT), serum alkaline phosphatase (ALP), total bilirubin
* Colonization with organisms associated with a more rapid decline in pulmonary status (for example, Burkholderia cenocepacia, Burkholderia dolosa, and Mycobacterium abscessus) at screening
* History of solid organ or hematological transplantation
* History of alcohol, medication or illicit drug abuse within 1 year before the first dose of study drug
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within 30 days before screening
* Any "non-CF-related" illness within 2 weeks before Day 1 (first dose of study drug). "Illness" was defined as an acute (serious or non-serious) condition (for example, gastroenteritis)
* Use of any inhibitors or inducers of cytochrome (CYP) P450 3A

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moss, MD, Principal Investigator — Stanford University
Locations (31):
- United States (29):
  - Birmingham, Alabama
  - Palo Alto, California
  - Hartford, Connecticut
  - Tampa, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
- United Kingdom (2):
  - Belfast
  - Edinburgh

REFERENCES:
- [Derived] Moss RB, Flume PA, Elborn JS, Cooke J, Rowe SM, McColley SA, Rubenstein RC, Higgins M; VX11-770-110 (KONDUCT) Study Group. Efficacy and safety of ivacaftor in patients with cystic fibrosis who have an Arg117His-CFTR mutation: a double-blind, randomised controlled trial. Lancet Respir Med. 2015 Jul;3(7):524-33. doi: 10.1016/S2213-2600(15)00201-5. Epub 2015 Jun 9. PMID 26070913

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 70 subjects were randomized, of which 1 subject discontinued the study prior to study drug administration. A total of 69 subjects started treatment.
Period: Overall Study
Arm/Group | Ivacaftor | Placebo
Started | 34 | 35
Completed | 32 | 35
Not Completed | 2 | 0
Not completed — Non-Compliance | 1 | 0
Not completed — Pregnancy (Self or Partner) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivacaftor | Placebo | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (16.57) | 32.7 (17.43) | 31.0 (16.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male subjects 18 years and older and female subjects 16 years and older. The Wang standard was used for male subjects aged 6 to 17 years and for female subjects aged 6 to 15 years.
Time Frame: Baseline, Week 24
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 34 | 35
percent predicted of FEV1 | 2.5724 (1.1532) | 0.4611 (1.1313)
Statistical Analysis 1: Comparison: Ivacaftor vs Placebo; Analysis was based on mixed effects model for repeated measures (MMRM) with dependent variable absolute change from baseline, with treatment group, visit and treatment by visit interaction as fixed effects, subject as random effect, and with adjustment for the continuous baseline value of age and percent predicted FEV1, using compound symmetry covariance matrix; Test type: Superiority or Other; p = 0.1979, Mixed Model Repeated Measures; Least squares (LS) Mean Difference = 2.1114, 95% CI 2-sided [-1.1305 to 5.3532]

2. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: Baseline, Week 24
Population: FAS included all randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 34 | 35
kg/m^2 | 0.4910 (0.6653) | 0.2284 (0.6504)
Statistical Analysis 1: Comparison: Ivacaftor vs Placebo; Analysis was based on linear mixed model with dependent variable BMI and treatment as a fixed effect, adjustment for baseline percent predicted FEV1, age and visit by treatment interaction was included as covariates and intercept, visit were included as random effects; Test type: Superiority or Other; p = 0.7780, Linear Mixed model — p-value for the treatment effect is from the slope of BMI (kg/m2) versus time (days); LS Mean difference = 0.2626, 95% CI 2-sided [-1.5698 to 2.0950]

3. Secondary Outcome: Change From Baseline in Sweat Chloride Through Week 24
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride.
Time Frame: Baseline, Week 24
Population: FAS included all randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo). Here, "Number of participants analyzed" signifies those subjects who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 32 | 35
millimole per liter (mmol/L) | -26.2771 (1.4584) | -2.3078 (1.3716)
Statistical Analysis 1: Comparison: Ivacaftor vs Placebo; Analysis was based on MMRM with dependent variable absolute change from baseline, with treatment group, visit and treatment by visit interaction as fixed effects, subject as random effect, and with adjustment for the continuous baseline value of age and percent predicted FEV1, and sweat chloride, using a compound symmetry covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; LS Mean difference = -23.9693, 95% CI 2-sided [-28.0094 to -19.9293]

4. Secondary Outcome: Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 24
Description: The CFQ-R is a validated subject-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 33 | 34
units on a scale | 7.5585 (2.2073) | -0.8289 (2.1569)
Statistical Analysis 1: Comparison: Ivacaftor vs Placebo; Analysis was based on MMRM with dependent variable absolute change from baseline, with treatment group, visit and treatment by visit interaction as fixed effects, subject as random effect, and with adjustment for the continuous baseline value of age and percent predicted FEV1, and CFQ-R respiratory domain score, using compound symmetry covariance matrix; Test type: Superiority or Other; p = 0.0091, Mixed Model Repeated Measures; LS Mean difference = 8.3874, 95% CI 2-sided [2.1658 to 14.6090]

5. Secondary Outcome: Time to First Pulmonary Exacerbation
Description: Number of events (pulmonary exacerbation) during the pre-specified time intervals were reported. A subject without an exacerbation before withdrawal from the study was considered censored at the time of withdrawal, and a subject without an exacerbation who completes the study period was considered censored at the end of the analysis period.
Time Frame: Day 0 to 15, Day 16 to 56, Day 57 to 112, Day 113 to 168
Population: FAS included all randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Measure: Number; unit: events
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 34 | 35
events
  Day 0 to 15 | 3 | 1
  Day 16 to 56 | 4 | 2
  Day 57 to 112 | 2 | 6
  Day 113 to 168 | 1 | 4
Statistical Analysis 1: Comparison: Ivacaftor vs Placebo; Test type: Superiority or Other; p = 0.8556, Cox Proportional Hazard Regression; Hazard Ratio (HR) = 0.928

6. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence, including clinically significant clinical laboratory assessments which occurs during course of study, whether it is considered related to study drug or not. SAE: medical event or condition, which falls into any of following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolonged hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, important medical event.
Time Frame: Baseline up to follow-up (3 to 4 weeks after last dose [last dose = Week 24])
Population: Safety Set included all subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Measure: Number; unit: participants
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 34 | 35
participants
  Subjects with any AEs | 32 | 35
  Subjects with SAEs | 4 | 6

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (3 to 4 weeks after last dose [last dose = Week 24])
Arm/Group | Ivacaftor | Placebo
Serious Adverse Events (participants affected / at risk) | 4/34 | 6/35
Other Adverse Events (participants affected / at risk) | 32/34 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (N=34) | Placebo (N=35)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 6
Cellulitis (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (N=34) | Placebo (N=35)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 11 | 13
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Sinusitis (Infections and infestations) | 2 | 5
Bacterial disease carrier (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 1 | 2
Acute sinusitis (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Scarlet fever (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 1
Palatal oedema (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 6
Fatigue (General disorders) | 2 | 2
Influenza like illness (General disorders) | 2 | 0
Pain (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Forced expiratory volume decreased (Investigations) | 3 | 2
Blood potassium increased (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1
Headache (Nervous system disorders) | 6 | 5
Dizziness (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Anal injury (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.